CLINICAL TRIAL: NCT05415865
Title: The Effect of Intravesical Lidocaine Solution Versus Placebo as Anesthesia Prior to Intravesical Injection of Onabotulinum Toxin A. A Randomized, Double-blind, Placebo Controlled Cross-over Study
Brief Title: The Effect of Local Anesthetic Solution in the Bladder Prior to Botox Injections in the Bladder
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Herlev and Gentofte Hospital (Other)
Collaborators: Region Hovedstadens Apotek (Other Government)
Responsible Party: Principal Investigator, Meryam El Issaoui, MD, PhD Student, Herlev and Gentofte Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: BTXA2021
Record Dates: First submitted 2022-06-08; First posted 2022-06-13 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Urge Incontinence; Overactive Bladder; Anesthesia, Local; Pain, Procedural; Urinary Tract Infections; Hematuria
Keywords: Urge incontinence; Anesthesia, Local; Botulinum Toxins, Type A; Overactive Bladder; Alkalinized Lidocaine; Double-blind Method; Visual Analog Scale; Administration, Intravesical
MeSH Terms: conditions — Urinary Incontinence, Urge; Urinary Bladder, Overactive; Pain, Procedural; Urinary Tract Infections; Hematuria

STUDY DESIGN:
Intervention Model Description: The study is a randomized, controlled, double-blinded, crossover study. The participants are their own control in the evaluation of the effect of intravesical alkalinized Lidocaine solution versus placebo as anesthesia prior to intravesical injection of onabotulinum toxin A. The chosen model is advantageous as a smaller sample size is needed, and error variance is reduced.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Region Hovedstadens Apotek, Herlev Hospital produces the Lidocaine solution and the matching placebo solution, performs the randomization, and packages the blinded dosing kits with the order of Lidocaine and placebo in a balanced design (50% Lidocaine at the first treatment). Participants will get consecutive randomization numbers, which specify the dosing kit. Neither the participant, the operator, or the healthcare professional interviewing the participant about her pain score know what solution the participant gets administered.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alkalinized Lidocaine, then Placebo (Active Comparator): Participants will have Lidocaine Hydrochloride 20 mg/ml, 20 ml and Sodium hydrogen carbonate 1 mmol/ml, 10 ml (ie a total of 30 ml) installed in the bladder for 15 minutes prior to the BTXA-injection procedure.
  When signing up for the next BTXA-injection with a wash out period of minimum three months, participants will have the matching placebo containing Sodium Chloride 9 g/L, 20 ml and Sodium Chloride 9 g/L, 10 ml, a total of 30 ml installed in the bladder for 15 minutes prior to the BTXA-injection procedure.
  Interventions: Combination Product: Alkalinized Lidocaine; Drug: Placebo Sodium Chloride 0.9% Inj
- Placebo, then Alkalinized Lidocaine (Active Comparator): Participants will have placebo containing Sodium Chloride 9 g/L, 20 ml and Sodium Chloride 9 g/L, 10 ml, a total of 30 ml installed in the bladder 15 minutes prior to the BTXA-injection procedure.
  When signing up for the next BTXA-injection with a wash out period of minimum three months, participants will have Lidocaine Hydrochloride 20 mg/ml, 20 ml and Sodium hydrogen carbonate 1 mmol/ml, 10 ml (ie a total of 30 ml) installed in the bladder for 15 minutes prior to the BTXA-injection procedure.
  Interventions: Combination Product: Alkalinized Lidocaine; Drug: Placebo Sodium Chloride 0.9% Inj

INTERVENTIONS:
Combination Product: Alkalinized Lidocaine — 20 ml of Lidocaine Hydrochloride and 10 ml of Sodium hydrogen carbonate will be pulled up and mixed in a syringe on site, and 30 ml mixed solution in total will afterwards be installed in the bladder with a catheter.
Drug: Placebo Sodium Chloride 0.9% Inj — 20 ml of Sodium Chloride 9 g/L and 10 ml of Sodium Chloride 9 g/L will be pulled up and mixed in a syringe on site, and 30 ml solution in total will afterwards be installed in the bladder with a catheter.

SUMMARY:
The purpose of this study is to investigate the effect of Lidocaine solution versus placebo (isotonic Sodium Chloride NaCl) disposed inside the urinary bladder as intravesical anesthesia prior to onabotulinum toxin A injections in the treatment of urgency urinary incontinence.

DETAILED DESCRIPTION:
The aim of the study is to investigate if bladder installed Lidocaine solution have an effect on reported pain during BTX-A injections compared to placebo.

The study participants will be recruited from the existing patient populations enrolled in the BTX-A program of the tertiary Urogynaecological Clinic of Herlev University Hospital.

The participants are randomized to:

1. Active drug: Lidocaine Hydrochloride and Sodium hydrogen carbonate
2. Placebo: Sodium Chloride

The study includes 5 study visits:

Visit 1:

* First treatment day
* Randomization
* Registration of pre-treatment pain relief medications: paracetamol, ibuprofen, or other medications. If pre-treatment pain relief is taken before first treatment, same pain relief should be taken before second treatment day (visit 4) in order to reduce bias
* Registration of antibiotic treatment: current antibiotic treatment or long-term prophylactic antibiotic for prevention of recurrent UTI The participant receives the active treatment or placebo, double-blinded
* The participant is asked to grade the intensity of pain according to VAS score immediately after, and when participant has been dressed after the BTX-A injections

Visit 2 (by telephone):

* Phone consultation 1 week after treatment:
* The participant's experience on the procedure on a 5-point ordinal scale: "1- very unsatisfied", "2- unsatisfied", "3- neither unsatisfied or satisfied", "4- satisfied", "5-very satisfied"

Side effects:

* Questions on symptoms of UTI: dysuria, cloudy urine, pollakiuria, nocturia
* Hematuria
* Inability to empty the bladder
* Other symptoms

(Visit 3:)

* The participant contacts the Clinic for next treatment approximately 6-12 months later
* Sponsor or investigator from the Urogynecological Clinic reach out for the participant asking on symptoms of UUI if the participant has not contacted the clinic within 12 months

Visit 4:

* Second treatment day
* The participant receives the opposite treatment, still double-blinded
* Registration of pre-treatment pain relief medications: paracetamol, ibuprofen, or other medications
* Registration of antibiotic treatment: current antibiotic treatment or long-term prophylactic antibiotic for prevention of recurrent UTI
* The participant is asked to grade the intensity of pain according to VAS score immediately after, and when participant has been dressed after the BTX-A injections

Visit 5(by telephone):

* Phone consultation 1 week after treatment:
* The participant's experience on the procedure on a 5-point scale: "1- very unsatisfied", "2- unsatisfied", "3- neither unsatisfied or satisfied", "4- satisfied", "5-very satisfied"

Side effects:

* Questions on symptoms of UTI: dysuria, cloudy urine, pollakiuria nocturia,
* Hematuria
* Inability to empty the bladder
* Other symptoms

ELIGIBILITY:
Inclusion criteria:

* Female, age ≥18 years
* Admitted to treatment with BTX-A injections at the Urogynecological Clinic at Herlev Hospital due to UUI
* Able to read and understand Danish
* The female accepts to receive BTX-A injections as an outpatient treatment without the option of receiving sedative drugs

Exclusion criteria:

* BTX-A allergy
* Neurological disorder that may affect bladder function (e.g. Multiple sclerosis or spinal cord inju-ry)
* Neurological disorder with neuromuscular transmission failure (i.e. Mystenia Gravis)
* Ongoing UTI or symptoms of UTI prior to treatment, assessed by principal investigator
* Any other bladder pathology at the time of cystoscopy if identified (includes trauma, stones, tu-mor)
* Pregnancy/breastfeeding women

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-09-12 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
100 mm Visual Analogue Scale (VAS) score | The participant is handed the VAS in paper form and asked to grade the intensity of pain according to the VAS by making a handwritten mark on the VAS immediately after the BTX-A injections
  The maximum pain score reported by using VAS

SECONDARY OUTCOMES:
Post-void residual requiring Clean Intermittent Catheterization (CIC) | Phone consultation one week after each treatment
  The participant is contacted after each treatment and asked about any inability to empty the bladder
Urinary tract infection (UTI) | Phone consultation one week after each treatment
  The participant is contacted after each treatment and asked about symptoms of UTI: Dysuria, cloudy urine, pollakiuria, nocturia
Hematuria | Phone consultation one week after each treatment
  The participant is contacted after each treatment and asked about blood in the urine
5-point rating scale | Phone consultation one week after each treatment
  The participant is contacted one week after every treatment and asked about the experience on the procedure. The participant's experience on the procedure on a 5-point ordinal scale: "1- very unsatis-fied", "2- unsatisfied", "3- neither unsatisfied or satisfied", "4- satisfied", "5-very satisfied"

CONTACTS AND LOCATIONS:
Overall Officials: Niels Klarskov, Prof,MD,DMSc, Study Director — Herlev and Gentofte Hospital, University of Copenhagen
Locations (1):
- Kvinde- og Bækkenbundssygdomme, klinik 1, Herlev, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haylen BT, de Ridder D, Freeman RM, Swift SE, Berghmans B, Lee J, Monga A, Petri E, Rizk DE, Sand PK, Schaer GN. An International Urogynecological Association (IUGA)/International Continence Society (ICS) joint report on the terminology for female pelvic floor dysfunction. Int Urogynecol J. 2010 Jan;21(1):5-26. doi: 10.1007/s00192-009-0976-9. Epub 2009 Nov 25. PMID 19937315
- [Background] Vaughan CP, Johnson TM 2nd, Ala-Lipasti MA, Cartwright R, Tammela TL, Taari K, Auvinen A, Tikkinen KA. The prevalence of clinically meaningful overactive bladder: bother and quality of life results from the population-based FINNO study. Eur Urol. 2011 Apr;59(4):629-36. doi: 10.1016/j.eururo.2011.01.031. Epub 2011 Jan 25. PMID 21306820
- [Background] Irwin DE, Milsom I, Kopp Z, Abrams P; EPIC Study Group. Symptom bother and health care-seeking behavior among individuals with overactive bladder. Eur Urol. 2008 May;53(5):1029-37. doi: 10.1016/j.eururo.2008.01.027. Epub 2008 Jan 16. PMID 18243515
- [Background] Nitti VW, Ginsberg D, Sievert KD, Sussman D, Radomski S, Sand P, De Ridder D, Jenkins B, Magyar A, Chapple C; 191622-096 Investigators. Durable Efficacy and Safety of Long-Term OnabotulinumtoxinA Treatment in Patients with Overactive Bladder Syndrome: Final Results of a 3.5-Year Study. J Urol. 2016 Sep;196(3):791-800. doi: 10.1016/j.juro.2016.03.146. Epub 2016 Mar 30. PMID 27038769
- [Background] Nambiar AK, Younis A, Khan ZA, Hildrup I, Emery SJ, Lucas MG. Alkalinized lidocaine versus lidocaine gel as local anesthesia prior to intra-vesical botulinum toxin (BoNTA) injections: A prospective, single center, randomized, double-blind, parallel group trial of efficacy and morbidity. Neurourol Urodyn. 2016 Apr;35(4):522-7. doi: 10.1002/nau.22750. Epub 2015 Mar 8. PMID 25754188
- [Background] Nickel JC, Moldwin R, Lee S, Davis EL, Henry RA, Wyllie MG. Intravesical alkalinized lidocaine (PSD597) offers sustained relief from symptoms of interstitial cystitis and painful bladder syndrome. BJU Int. 2009 Apr;103(7):910-8. doi: 10.1111/j.1464-410X.2008.08162.x. Epub 2008 Nov 13. PMID 19021619
- [Background] Henry R, Patterson L, Avery N, Tanzola R, Tod D, Hunter D, Nickel JC, Morales A. Absorption of alkalized intravesical lidocaine in normal and inflamed bladders: a simple method for improving bladder anesthesia. J Urol. 2001 Jun;165(6 Pt 1):1900-3. doi: 10.1097/00005392-200106000-00014. PMID 11371877
- [Background] Narahashi T, Frazier T, Yamada M. The site of action and active form of local anesthetics. I. Theory and pH experiments with tertiary compounds. J Pharmacol Exp Ther. 1970 Jan;171(1):32-44. No abstract available. PMID 5410936
- [Background] Henry RA, Patterson L, Nickel C, Morales A. Alkalinized intravesical lidocaine to treat interstitial cystitis: absorption kinetics in normal and interstitial cystitis bladders. Urology. 2001 Jun;57(6 Suppl 1):119. doi: 10.1016/s0090-4295(01)01069-x. No abstract available. PMID 11378101
- [Background] Yanagi H, Sankawa H, Saito H, Iikura Y. Effect of lidocaine on histamine release and Ca2+ mobilization from mast cells and basophils. Acta Anaesthesiol Scand. 1996 Oct;40(9):1138-44. doi: 10.1111/j.1399-6576.1996.tb05577.x. PMID 8933856
- [Background] Pereira E Silva R, Ponte C, Lopes F, Palma Dos Reis J. Alkalinized lidocaine solution as a first-line local anesthesia protocol for intradetrusor injection of onabotulinum toxin A: Results from a double-blinded randomized controlled trial. Neurourol Urodyn. 2020 Nov;39(8):2471-2479. doi: 10.1002/nau.24519. Epub 2020 Sep 21. PMID 32956506
- [Background] Nitti VW, Dmochowski R, Herschorn S, Sand P, Thompson C, Nardo C, Yan X, Haag-Molkenteller C; EMBARK Study Group. OnabotulinumtoxinA for the treatment of patients with overactive bladder and urinary incontinence: results of a phase 3, randomized, placebo controlled trial. J Urol. 2013 Jun;189(6):2186-93. doi: 10.1016/j.juro.2012.12.022. Epub 2012 Dec 14. PMID 23246476
- [Background] Duthie JB, Vincent M, Herbison GP, Wilson DI, Wilson D. Botulinum toxin injections for adults with overactive bladder syndrome. Cochrane Database Syst Rev. 2011 Dec 7;2011(12):CD005493. doi: 10.1002/14651858.CD005493.pub3. PMID 22161392
- [Background] Dmochowski R, Chapple C, Nitti VW, Chancellor M, Everaert K, Thompson C, Daniell G, Zhou J, Haag-Molkenteller C. Efficacy and safety of onabotulinumtoxinA for idiopathic overactive bladder: a double-blind, placebo controlled, randomized, dose ranging trial. J Urol. 2010 Dec;184(6):2416-22. doi: 10.1016/j.juro.2010.08.021. Epub 2010 Oct 16. PMID 20952013
- [Background] Cote TR, Mohan AK, Polder JA, Walton MK, Braun MM. Botulinum toxin type A injections: adverse events reported to the US Food and Drug Administration in therapeutic and cosmetic cases. J Am Acad Dermatol. 2005 Sep;53(3):407-15. doi: 10.1016/j.jaad.2005.06.011. PMID 16112345
- [Background] Thrasher JB, Peterson NE, Donatucci CF. Lidocaine as a topical anesthetic for bladder biopsies. J Urol. 1991 Jun;145(6):1209-10. doi: 10.1016/s0022-5347(17)38577-4. PMID 2033694
- [Background] Thrasher JB, Kreder KJ, Peterson NE, Donatucci CF. Lidocaine as topical anesthesia for bladder mappings and cold-cup biopsies. J Urol. 1993 Aug;150(2 Pt 1):335-6. doi: 10.1016/s0022-5347(17)35477-0. PMID 8326556
- [Background] Birch BR, Miller RA. Absorption characteristics of lignocaine following intravesical instillation. Scand J Urol Nephrol. 1994 Dec;28(4):359-64. doi: 10.3109/00365599409180513. PMID 7886411
- [Derived] El Issaoui M, Elmelund M, Klarskov N. Alkalinised lidocaine as an anaesthetic before onabotulinumtoxinA injections. a randomised trial. BJU Int. 2025 Apr;135(4):638-647. doi: 10.1111/bju.16647. Epub 2025 Jan 11. PMID 39797697
- See also: Abrams P, Cardozo, L, Wagg, A, Wein, A. (Eds) Incontinence 6th Edition. International Continence Society, Bristol UK,: ICI-ICS.; 2017 — https://www.ics.org/education/icspublications/icibooks/6thicibook
- See also: Incontinence. International Consultation on Incontinence: ICUD; 2017 — https://www.ics.org/education/icspublications/icibooks/6thicibook